CLINICAL TRIAL: NCT06324903
Title: Role of Echocardiography in Optimization of Cardiac Catheterization Performance in Children With Congenital Heart Disease
Brief Title: Role of Echocardiography in Optimization of Cardiac Catheterization in Children With Congenital Heart Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Abdelmonem Abdelgalil Mohamed, principle investigator, Assiut University
Other Study IDs: echo cath CHD
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: echocardiography and percutaneous cardiac catheterization — pre- cardiac catheterization, intraprocedural and post-catheterization echocardiography.

SUMMARY:
Delineate and evaluate the role of echocardiography in children with congenital heart disease undergoing cardiac catheterization in the pediatric cardiology unit of Assiut university hospitals.

1. To improve diagnostic accuracy by creating a systematic approach for image acquisition and interpretation across different procedural timepoints.
2. To promote consistent hemodynamic evaluations to reliably assess cardiac function and blood flow.
3. To enable optimized procedural planning and intraprocedural guidance via comprehensive delineation of anatomy and pathophysiology.
4. To facilitate standardized longitudinal monitoring after interventions to evaluate outcomes and detect complications.

DETAILED DESCRIPTION:
Congenital heart disease is estimated to affect approximately 1% of live births, underscoring the profound impact of this set of cardiac malformations . Echocardiography serves as the cornerstone imaging modality utilized in all aspects of care in this patient population - from initial diagnosis, to informing surgical and transcatheter interventions, to longitudinal surveillance . Recent decades have witnessed major advancements in the catheter-based treatment of Congenital heart disease , sparing patients from more invasive open-heart procedures in select cases . Transcatheter closure of defects such as atrial septal defects , ventricular septal defects and patent ductus arteriosus have become mainstream interventions . However, the complexity of Congenital heart disease anatomy necessitates meticulous procedural planning and guidance to achieve optimal outcomes following these catheterizations .

Importance of Standardized Echocardiography Protocols Echocardiography is invaluable before, during and after transcatheter interventions in patients with congenital heart disease. Precise delineation of anatomy facilitates appropriate procedure selection and planning - including choice of access, devices, and imaging guidance . Intraprocedural transesophageal echocardiography offers real-time visualization for device positioning and deployment as well as identification of complications . Post-intervention surveillance detects residual lesions, enables assessment of ventricular function and valvular regurgitation, and monitors for complications such as thrombosis or device erosion .

Despite extensive guidelines on the echocardiographic assessment of congenital heart disease, substantial inter-institutional variability persists in imaging for catheter-based procedures . Standardized protocols have demonstrated improvements in accuracy, consistency, and quality . However, adoption of such protocols is lagging. This gap highlights the pressing need for evidence-based protocols to optimize echocardiography practices.

This proposed protocol focuses on pre-catheterization, intraprocedural and post-catheterization transthoracic echocardiography and transesophageal echocardiography for common interventions - atrial septal defects closure, ventricular septal defects closure and patent ductus arteriosus closure. It provides comprehensive recommendations on essential views, measurements, and documentation. The protocol allows modularity to adapt components across different interventions. Wider adoption has the potential to substantially improve consistency, accuracy, patient safety and quality. Further studies are imperative to demonstrate the impact of implementing such standardized protocols. This initiative represents an important step towards advancing care for pediatric catheterizations.

ELIGIBILITY:
Inclusion Criteria:

* All infants and children from 1month to 18 years old with congenital cardiac defects indicated for cardiac catheterization

Exclusion Criteria:

* • Patients with complex cardiac disease,

  * Patients with a history of renal disease,
  * Patient who are less than 1 month,
  * Parental refusal to participate in the research.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Infants and children age from 1 month to 18 years old. Hospitalized patients in pediatric cardiology unit, Assiut University Hospitals, who are prepared for cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
congenital heart defect dimensions in mm, | 2 DAYS
  congenital heart defect dimensions in mm which are patent ductus arteriosus (PDA), ventricular septal defect (VSD), atrial septal defect (ASD) dimensions in (mm) millimeter.
  comparing pre-catheter and intra-catheter procedure measurement measuring by transthoracic echocardiography 24 hours pre-catheter then intra-catheter by transesophageal echocardiography and transcatheter angiography.
pressure gradient in mmHg across valve | 2 DAYS
  pressure gradient in mmHg which are valvular pulmonary stenosis (VPS) pressure gradient in mmHg. pulmonary hypertension measured in mmHg. comparing pre-catheter and intra-catheter procedure measurement measuring by transthoracic echocardiography 24 hours pre-catheter then intra-catheter by transesophageal echocardiography and transcatheter angiography.

SECONDARY OUTCOMES:
cardiac function by measuring fraction shortening (FS) % in percent | 6 months
  echocardiography measurements of cardiac systolic function for 24 hours pre-catheterization studies, for 48 hours post-catheterization studies and on 6 months follow up ( LVEDD in mm, LVESD in mm, , FS in % ( Fractional shortening (FS) = LVEDD-LVESD/LVESD ×100 )
cardiac function TAPSV in cm/sec | 6 months
  cardiac function of right side of the heart TAPSV in cm/sec, echocardiography tissue doppler measurements of cardiac systolic function for 24 hours pre-catheterization studies, for 48 hours post-catheterization studies and on 6 months follow up TAPSV in cm/sec.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Background] Sachdeva R, Valente AM, Armstrong AK, Cook SC, Han BK, Lopez L, Lui GK, Pickard SS, Powell AJ, Bhave NM, Sachdeva R, Valente AM, Pickard SS, Baffa JM, Banka P, Cohen SB, Glickstein JS, Kanter JP, Kanter RJ, Kim YY, Kipps AK, Latson LA, Lin JP, Parra DA, Rodriguez FH 3rd, Saarel EV, Srivastava S, Stephenson EA, Stout KK, Zaidi AN. ACC/AHA/ASE/HRS/ISACHD/SCAI/SCCT/SCMR/SOPE 2020 Appropriate Use Criteria for Multimodality Imaging During the Follow-Up Care of Patients With Congenital Heart Disease: A Report of the American College of Cardiology Solution Set Oversight Committee and Appropriate Use Criteria Task Force, American Heart Association, American Society of Echocardiography, Heart Rhythm Society, International Society for Adult Congenital Heart Disease, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, Society for Cardiovascular Magnetic Resonance, and Society of Pediatric Echocardiography. J Am Coll Cardiol. 2020 Feb 18;75(6):657-703. doi: 10.1016/j.jacc.2019.10.002. Epub 2020 Jan 6. No abstract available. PMID 31918898
- [Background] Ramlawi B. The Era of Catheter-Based and Minimally Invasive Cardiac Surgery. Methodist Debakey Cardiovasc J. 2016 Jan-Mar;12(1):3. doi: 10.14797/mdcj-12-1-3. No abstract available. PMID 27127554
- [Background] Turner ME, Bouhout I, Petit CJ, Kalfa D. Transcatheter Closure of Atrial and Ventricular Septal Defects: JACC Focus Seminar. J Am Coll Cardiol. 2022 Jun 7;79(22):2247-2258. doi: 10.1016/j.jacc.2021.08.082. PMID 35654496
- [Background] Divekar AA, Arar YM, Clark S, Tandon A, Zellers TM, Veeram Reddy SR. Transcatheter Device Therapy and the Integration of Advanced Imaging in Congenital Heart Disease. Children (Basel). 2022 Apr 2;9(4):497. doi: 10.3390/children9040497. PMID 35455541
- [Background] Avesani M, Kang SL, Jalal Z, Thambo JB, Iriart X. Renaissance of Cardiac Imaging to Assist Percutaneous Interventions in Congenital Heart Diseases:The Role of Three-Dimensional Echocardiography and Multimodality Imaging. Front Pediatr. 2022 May 19;10:894472. doi: 10.3389/fped.2022.894472. eCollection 2022. PMID 35664875
- [Background] Kenny D. Interventional Cardiology for Congenital Heart Disease. Korean Circ J. 2018 May;48(5):350-364. doi: 10.4070/kcj.2018.0064. Epub 2018 Mar 29. PMID 29671282
- [Background] Maragiannis D, Little SH. Interventional imaging: the role of echocardiography. Methodist Debakey Cardiovasc J. 2014 Jul-Sep;10(3):172-7. doi: 10.14797/mdcj-10-3-172. PMID 25574345
- [Background] Zhang X, Gosnell J, Nainamalai V, Page S, Huang S, Haw M, Peng B, Vettukattil J, Jiang J. Advances in TEE-Centric Intraprocedural Multimodal Image Guidance for Congenital and Structural Heart Disease. Diagnostics (Basel). 2023 Sep 18;13(18):2981. doi: 10.3390/diagnostics13182981. PMID 37761348
- [Background] Ludomirsky A. The use of echocardiography in pediatric interventional cardiac catheterization procedures. J Interv Cardiol. 1995 Oct;8(5):569-78. doi: 10.1111/j.1540-8183.1995.tb00584.x. PMID 10159521
- [Background] Little SH, Rigolin VH, Garcia-Sayan E, Hahn RT, Hung J, Mackensen GB, Mankad S, Quader N, Saric M. Recommendations for Special Competency in Echocardiographic Guidance of Structural Heart Disease Interventions: From the American Society of Echocardiography. J Am Soc Echocardiogr. 2023 Apr;36(4):350-365. doi: 10.1016/j.echo.2023.01.014. Epub 2023 Feb 24. PMID 36841670
- [Background] Broder MS, Gibbs SN, Yermilov I. An Adaptation of the RAND/UCLA Modified Delphi Panel Method in the Time of COVID-19. J Healthc Leadersh. 2022 May 20;14:63-70. doi: 10.2147/JHL.S352500. eCollection 2022. PMID 35634010
- [Background] Sharma AK, Agarwal A, Sinha SK, Razi MM, Pandey U, Shukla P, Thakur R, Verma CM, Bansal RK, Krishna V. An echocardiographic evaluation to determine the immediate and short-term changes in biventricular systolic and diastolic functions after PDA device closure-an observational analytical prospective study (echo- PDA study). Indian Heart J. 2021 Sep-Oct;73(5):617-621. doi: 10.1016/j.ihj.2021.06.017. Epub 2021 Jul 6. PMID 34627579
- [Background] Hou M, Qian W, Wang B, Zhou W, Zhang J, Ding Y, Xu Q, Huang J, Shen J, Cao L, Lv H, Sun L. Echocardiographic Prediction of Left Ventricular Dysfunction After Transcatheter Patent Ductus Arteriosus Closure in Children. Front Pediatr. 2019 Oct 15;7:409. doi: 10.3389/fped.2019.00409. eCollection 2019. PMID 31681709